CLINICAL TRIAL: NCT07238465
Title: Dysautonomia InVestigation in Individuals With Down SyndromE: DIVE Study
Brief Title: Exploring Sympathetic Nervous System Function in Individuals With Down Syndrome
Acronym: DIVE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Linda Crnic Institute for Down Syndrome (Unknown); GLOBAL Down Syndrome Foundation (Unknown); University of Colorado Colorado Clinical and Translational Sciences Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 25-0503; T32AG000279 (NIH)
Record Dates: First submitted 2025-10-22; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Down Syndrome; Autonomic Dysfunction
Keywords: Cold Stress; Pain Responses; Fear; Exercise; Blood Pressure; Heart Rate; Caffeine; 12-Hour Fast; Catecholamines; Epinephrine; Norepinephrine; Dopamine
MeSH Terms: conditions — Down Syndrome; Primary Dysautonomias; Motor Activity | interventions — Cold-Shock Response; Caffeine; Coffee; Hig1 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Down syndrome (Experimental): The investigators will be recruiting participants between the ages of 18-50 for the study investigating responses to six sympathetic stressors compared to age and sex matched individuals without Down syndrome.
  Interventions: Other: Fear Response; Other: Cold Stress; Other: Pain Response; Other: Caffeine; Other: 12-Hour Fast; Other: Maximal Dynamic Exercise
- Individuals without Down syndrome (Experimental): The investigators will be recruiting individuals without Down syndrome between the ages of 18-50 to serve as the comparisons for individuals with Down syndrome across the six sympathetic stressors.
  Interventions: Other: Fear Response; Other: Cold Stress; Other: Pain Response; Other: Caffeine; Other: 12-Hour Fast; Other: Maximal Dynamic Exercise

INTERVENTIONS:
Other: Fear Response — Fear triggers the sympathetic nervous system, known as the 'fight-or-flight' response, which prepares the body to respond to a perceived threat by increasing heart rate, blood pressure, and releasing catecholamines. These measurements will be taken to examine the cardiovascular physiology of how individuals with DS will respond during a scary simulation.
  The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed during a fear simulation using virtual reality goggles in individuals with Down syndrome, who have proposed autonomic dysfunction. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: Physiological Fear Response; Virtual Reality Simulation
Other: Cold Stress — Cold triggers the sympathetic nervous system, known as the 'fight-or-flight' response, which prepares the body to respond to a perceived threat by increasing heart rate, blood pressure, and releasing catecholamines. These measurements will be taken to examine how individuals with DS will respond during a cold stress test.
  The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed during a cold stress test in individuals with Down syndrome, who have proposed autonomic dysfunction. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: Cold Pressor Test; Cold Water
Other: Pain Response — Pain triggers the sympathetic nervous system, known as the 'fight-or-flight' response, which prepares the body to respond to the perceived threat (i.e., hurt) by increasing heart rate, blood pressure, and releasing catecholamines. These measurements will be taken to examine how individuals with DS will respond during application of a painful patch.
  The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed during application of a pain patch in individuals with Down syndrome, who have proposed autonomic dysfunction. This pain patch is similar to what someone would buy at the drug store for sore muscles. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: Capsaicin Patch
Other: Caffeine — Caffeine acts as a stimulant to the sympathetic nervous system leading to an increase in blood pressure, heart rate, and release of catecholamines.
  The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed following ingestion of a caffeine pill (similar to ~2 cups of coffee) in individuals with Down syndrome, who have proposed autonomic dysfunction. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: Caffeine Pill; Coffee
Other: 12-Hour Fast — Fasting-induced hypoglycemia triggers a 'fight-or-flight' response as the body attempts to raise low blood glucose levels to bring them back to 'normal'. These measurements will be taken to examine how individuals with DS will respond following a 12-hour abstinence from food, inducing low blood sugar.
  The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed following a 12-hour fast in individuals with Down syndrome, who have proposed autonomic dysfunction. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: Low Blood Sugar; Hypoglycemia
Other: Maximal Dynamic Exercise — The investigators are looking at how plasma catecholamines (i.e., Epinephrine, Norepinephrine, and Dopamine), blood pressure, and heart rate are expressed during a treadmill maximal exercise test in individuals with Down syndrome, who have proposed autonomic dysfunction. This study will compare responses among individuals with Down syndrome to a control group without Down syndrome.
  Other Names: VO2peak; Treadmill Exercise

SUMMARY:
Down syndrome (DS), the most common genetic cause of intellectual disability, is associated with widespread organ dysfunction, including abnormalities in the autonomic nervous system (ANS). The ANS regulates critical functions such as heart rate (HR) and blood pressure (BP), both essential for maintaining homeostasis and supporting physical activity. Individuals with DS often exhibit blunted HR responses to exercise-typically ~30 beats per minute below expected levels-suggesting reduced sympathetic nervous system (SNS) activity. The SNS governs rapid changes in HR and BP during stress by releasing catecholamines: epinephrine (from the adrenal medulla) and norepinephrine (from sympathetic nerve endings). Despite its importance, SNS function has not been comprehensively assessed among individuals with DS.

This study addresses a critical knowledge gap by evaluating SNS responses to physiological stressors in individuals with DS. The investigators will measure beat-to-beat HR and BP, along with plasma catecholamine levels, in response to sympathetic activation, comparing individuals with DS to age- and sex-matched controls. Understanding the mechanisms of SNS dysfunction in DS is vital, as it likely underlies reduced exercise capacity and contributes to broader clinical challenges. These insights may guide targeted interventions to improve cardiovascular function, physical capacity, and overall quality of life in this understudied population.

DETAILED DESCRIPTION:
Evolution has equipped each species with instinctual defense mechanisms to cope with environmental stressors, ensuring survival. Many of these mechanisms are driven by activation of the sympathetic nervous system (SNS), which orchestrates the "fight or flight" response. Systemic SNS activation extends across all organ systems, triggering the release of catecholamines to elevate heart rate (HR) and increase blood pressure (BP) to meet the heightened metabolic demands of the stressor and ensure the delivery of oxygen-rich blood to active tissues. Exercise, a potent sympathoexcitatory stressor, poses a major challenge to the oxygen transport system, requiring coordinated organ system function to increase both HR and BP. Dysregulated SNS activation can impair oxygen delivery, leading to reduced work capacity, quality of life, and is an independent predictor of morbidity and premature mortality. Therefore, experimental approaches to understand SNS activation in populations with reduced work capacity and premature morbidity, mortality is of upmost importance for improving health outcomes and quality of life on a population level.

Down syndrome (DS) is the most common chromosomal abnormality in the human population, with widespread effects across numerous tissues and organ systems, including accelerated biological aging. Individuals with DS exhibit reduced work capacity, with maximal HRs ~30 beats below normal, and face higher rates of premature morbidity and mortality than the general population. Notably, individuals with DS demonstrate blunted catecholamine response to the sympathetic stressor of maximal exercise, suggesting diminished SNS activation. Recent literature from this PI suggests altered peripheral blood flow and BP regulation among individuals with DS during large muscle mass exercise which immolates walking, or running- critical for survival. These findings align with recent evidence of hypoxic signaling, elevated heme metabolism, and stress erythropoiesis across the lifespan in this population. Together, these data suggest that impaired oxygen delivery, potentially linked to SNS dysregulation, may be more widespread in DS than previously recognized.

However, the role of SNS activation in the context of daily stressors which elevate both HR and BP, remains unclear. Understanding the mechanisms underlying SNS dysfunction in DS is crucial, as it likely contributes to many clinical and developmental challenges, including the underlying reduced work capacity and suggested autonomic dysfunction observed in this population. Addressing this gap may enable targeted therapies to enhance survival, longevity, and quality of life for individuals with DS. The investigators aim to systematically evaluate SNS activation through six stressors which mimic common stressors faced to any individual over the course of a day or lifespan. Through evaluation of plasma catecholamines, the investigators hope to elucidate the mechanisms and impact of catecholamine responses in individuals with DS compared typical responses observed among individuals without DS.

Aim 1. Characterize the catecholamine response to physiological stressors among individuals with DS. The investigators will assess SNS responses in individuals with DS and age- and sex-matched controls. Beat-to-beat HR and BP, along with plasma catecholamine levels will be collected in response to the following sympathetic stressors: A) Cold Stress, B) Fear (i.e., virtual reality), C) Pain (i.e., capsicum patch), D) Caffeine, E) 12-Hour Fast, and F) Maximal Dynamic Exercise (VO2peak). Metabolomics and proteomics will be performed on the plasma samples and these efforts will help define the manifestations of hormonal SNS dysfunction in individuals with DS.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 yrs old and apparently healthy individuals
* Ability to understand the study and give assent to participate
* Has a study partner who can attend all visits for the individuals with DS, and answer questionnaires, provide consent when necessary
* Corrected or non-existent congenital heart disease
* Euthyroid or on stable thyroid medication dose for at least 6 months
* Free from cardiovascular, pulmonary, inflammatory, or metabolic disease in the past 6 months that would prevent participation in study procedures
* BMI <45kg/m2
* Ability to tolerate repeated blood draws / catheter placement

Exclusion Criteria:

* Hypertension (resting systolic blood pressure [SBP] ≥140 and/or diastolic blood pressure [DBP] ≥90 mmHg) this includes those on medications to treat hypertension
* Hypotension (resting BP of <90/60 mmHg)
* Cancer in the last six months
* Any heart-rate-altering medications or any other medication that may modify metabolic responses
* Self-reported diabetes or use of glucose-lowering medication
* Tobacco products, including vaping, or marijuana use
* Currently pregnant
* Post-menopausal women

Specific Exclusion Criteria for Certain Stressors:

* Orthopedic limitations that would prohibit exercise or movement for exercise
* Fracture of limb to be immersed for CPT
* Open cut or sore on hand to be immersed for CPT
* Raynaud's syndrome for CPT
* Chronic caffeine drinkers for caffeine stressor (consumption of caffeine in the last 7 days)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Seated Baseline Concentration of Plasma Catecholamines | Seated baseline blood draw, prior to stressors
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Concentration of Plasma Catecholamines During Cold Pressor Test | During the cold stress test, around or up to 5 minutes
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Baseline Standing Concentration of Plasma Catecholamines | Standing baseline blood draws, prior to fear simulation
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
First Fear Simulation, Concentration of Plasma Catecholamines | During the first virtual reality fear stressor, around 5 minutes
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Second Fear Simulation, Concentration of Plasma Catecholamines | During the second fear simulation, around 15 minutes into the test
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
First Minute of Pain Patch, Concentration of Plasma Catecholamines | Blood draw will take place within 1-minute of the application of the pain patch.
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
15 Minutes into Pain Patch Application, Concentration of Plasma Catecholamines | Blood draw will occur about 15 minutes after the application of the pain patch.
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
12-Hour Fast, Concentration of Plasma Catecholamines | Blood draw will occur following a 12-hour fast inducing hypoglycemia
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Seated Baseline Blood Draw, Concentration of Plasma Catecholamines | Blood draw will occur prior to ingestion of caffeine pill
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
30 Minutes Following Ingestion of Caffeine Pill(s), Concentration of Plasma Catecholamines | Blood draw will occur around 30 minutes following participant ingestion of caffeine pill(s)
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
60 Minutes Following Ingestion of Caffeine Pill(s), Concentration of Plasma Catecholamines | Blood draw will occur around 60 minutes following participant ingestion of caffeine pill(s)
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Baseline Standing Concentration of Plasma Catecholamines Prior to Maximal Exercise Test | Standing baseline blood draw, prior to maximal exercise test
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Standing Concentration of Plasma Catecholamines at End of Maximal Exercise Test | This blood draw will occur at the very end or immediately following the maximal exercise test on the treadmill
  Investigators will use metabolomic techniques to quantify plasma concentrations of epinephrine, norepinephrine, and dopamine in all participants before, during (in some stressors), and after the six stressor tests. These metabolites will provide insight into sympathetic nervous system activation in individuals with Down syndrome compared to those without Down syndrome.
Seated Baseline Heart Rate, Prior to Cold Pressor Test | Resting seated baseline, prior to cold pressor test, up to or around 5 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during (in some stressors), and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate Collected During Cold Pressor Test | Collected throughout the Cold Pressor Test, around 6 minutes in total
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Standing Baseline Heart Rate, Prior to Fear Simulations | Standing baseline, prior to fear simulations, up to or around 5 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, First Fear Simulation | Continuous heart rate will be collected during the first fear simulation, which will last around or up to 10 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, First Calming Simulation | Continuous heart rate will be recorded during the first calming simulation, which will follow the first fear simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Second Fear Simulation | Continuous heart rate will be recorded during the second fear simulation, which will follow the first calming simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Second Calming Simulation | Continuous heart rate will be recorded during the second calming simulation, which will follow the second fear simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Baseline Prior to Pain Patch | Baseline seated heart rate recordings will occur prior to application of pain patch, up to or around 5 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, During Pain Patch | Continuous heart rate will be recorded following the application of the capsaicin pain patch, up to or around 15 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Baseline 12-Hour Fast | Resting baseline will be recorded prior (and on a separate day from) the 12-hour fast, up to or around 5 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, 12-Hour Fast | Seated heart rate recordings will occur following a 12-hour fast, up to or around 15 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Seated Baseline, Caffeine Consumption | Resting baseline heart rate will be recording prior to caffeine consumption, up to or around 5 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Following Caffeine Consumption | Continuous heart rate recordings will occur immediately following caffeine consumption, up to or around 60 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Baseline Prior to Maximal Exercise Test | Baseline heart rate recordings will occur prior to the maximal exercise test, up to or around 5 minutes.
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Heart Rate, Maximal Exercise Test | Continuous heart rate recordings will take place throughout the maximal aerobic exercise test on the treadmill, up to or around 20 minutes
  Investigators will collect beat-to-beat heart rate recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Seated Baseline Blood Pressure, Prior to Cold Pressor Test | Resting seated baseline, prior to cold pressor test, up to or around 5 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure Collected During Cold Pressor Test | Collected throughout the Cold Pressor Test, around 6 minutes in total
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Standing Baseline Blood Pressure, Prior to Fear Simulations | Standing baseline, prior to fear simulations, up to or around 5 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, First Fear Simulation | Continuous blood pressure will be recorded during the first fear simulation, which will last up to or around 10 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, First Calming Simulation | Continuous blood pressure will be recorded during the first calming simulation, which will follow the first fear simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Second Fear Simulation | Continuous blood pressure will be recorded during the second fear simulation, which will follow the first calming simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Second Calming Simulation | Continuous blood pressure will be recorded during the second calming simulation, which will follow the second fear simulation and will last up to or around 10 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Baseline Prior to Pain Patch | Baseline seated blood pressure recordings will occur prior to application of pain patch, up to or around 5 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, During Pain Patch | Continuous blood pressure will be recorded following the application of the capsaicin pain patch, up to or around 15 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Baseline 12-Hour Fast | Resting baseline will be recorded prior (and on a separate day from) the 12-hour fast, up to or around 5 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, 12-Hour Fast | Seated blood pressure recordings will occur following a 12-hour fast, up to or around 15 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Seated Baseline, Caffeine Consumption | Resting baseline blood pressure will be recording prior to caffeine consumption, up to or around 5 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Following Caffeine Consumption | Continuous blood pressure recordings will occur immediately following caffeine consumption, up to or around 60 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Baseline Prior to Maximal Exercise Test | Baseline blood pressure recordings will occur prior to the maximal exercise test, up to or around 5 minutes.
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.
Blood Pressure, Maximal Exercise Test | Continuous blood pressure recordings will take place throughout the maximal aerobic exercise test on the treadmill, up to or around 20 minutes
  Investigators will collect beat-to-beat blood pressure recordings in all participants before, during, and after the six stressor tests. These cardiovascular perturbations will provide insight into sympathetic nervous system modulation in individuals with Down syndrome compared to those without Down syndrome.

SECONDARY OUTCOMES:
Facial Affective Scale Score, Baseline Assessment | Baseline Assessment of Facial Affective Scale, this will occur prior to any stressors.
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score. This will take up to or around approximately 5 minutes to complete.
Facial Affective Scale Score, Cold Pressor Test, 1.5 Minutes | Assessment occurs around or up to 90 seconds (1.5 minutes) into cold water immersion
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Facial Affective Scale Score, Cold Pressor Test, Finale | Assessment occurs immediately following or during the last minute of the Cold Pressor Test, up to or around 6 minutes following placement of arm into cold
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Facial Affective Scale Score, During Pain Response, 1-Minute | Assessment will take place approximately 1-minute following administration of the pain patch
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Facial Affective Scale Score, Pain Response, 5 Minutes | Up to or around 5 minutes into pain patch
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Facial Affective Scale Score, Pain Response, 10 Minutes | Up to or around 10 minutes into pain patch application
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Facial Affective Scale Score, Pain Response, 15 Minutes | Up to or around 15 minutes following the application of the pain patch
  Investigators will use the validated 'Facial Affective Scale', which uses a series of nine drawn faces showing various degrees of emotional distress to help participants assess their emotional state. The nine faces represent a range of negative to positive affect, and each face having a specific value between 0.04 (maximum positive affect) and 0.97 (maximum negative affect). The chosen face's corresponding value is the Facial Affective Score.
Blood Glucose, Baseline Without 12-Hour Fast | Baseline without fast, Prior to 12-Hour fast condition to confirm low blood sugars
  Blood glucose measurements will be taken via a small capillary blood sample using a commercially available spring-loaded lancet. This will help to confirm the presence of low blood sugars among the participants for the 12-Hour Fast stressor.
Blood Glucose, 12-Hour Fast | Measurement will be conducted prior to the 12-Hour fast condition to confirm low blood sugars
  Blood glucose measurements will be taken via a small capillary blood sample using a commercially available spring-loaded lancet. This will help to confirm the presence of low blood sugars among the participants for the 12-Hour Fast stressor.

CONTACTS AND LOCATIONS:
Locations (1):
- Linda Crnic Institute for Down Syndrome, University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No